CLINICAL TRIAL: NCT04769310
Title: Advanced Cardiac Imaging To Predict Embolic Stroke On Brain MRI: A Pilot Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-2151
Record Dates: First submitted 2021-02-19; First posted 2021-02-24 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation; Stroke; Stroke, Cardiovascular; Vascular Cognitive Impairment; Strokes Thrombotic; Stroke, Ischemic
Keywords: Magnetic Resonance Imaging; Cardiac Magnetic Resonance Imaging; Brain infarcts; Left atrial; Left atrial appendage; Non invasive cardiac imaging
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Myocardial Infarction; Thrombotic Stroke; Ischemic Stroke; Brain Infarction

STUDY DESIGN:
Intervention Model Description: All patients will undergo a CMR to evaluate for LA and LAA high-risk features on either a 1.5 or 3 Tesla clinical MR scanner. CMR protocol will include Cine MRI, contrast-enhanced (CE) MR Angiography (MRA), time-resolved 2D phase-contrast (PC) MRI, and 3D late gadolinium enhancement (LGE) involving gadolinium injection. Gadolinium is a contrast product that helps define areas of fibrosis in the LA.
  Brain MRI will be used for the detection of embolic infarcts assessed on high-resolution brain MRI acquisitions. The high-resolution brain MRI with no contrast will include the following sequences for most accurate assessment of embolic lesions: 3D T1 Magnetization Prepared Rapid Acquisition Gradient Echo (MPRAGE), 3D fluid attenuated inversion recovery (FLAIR), diffusion weighted imaging (DWI), apparent diffusion coefficient maps (ADC), and susceptibility weighted imaging (SWI).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patient arm (Other): All patients will undergo a CMR to evaluate for LA and LAA high-risk features on either a 1.5 or 3 Tesla clinical MR scanner. Gadolinium injection will be administered. Gadolinium is a contrast product that helps define areas of fibrosis in the LA.
  High-resolution brain MRI with no contrast will include the following sequences for most accurate assessment of embolic lesions: 3D T1 MPRAGE, 3D FLAIR, DWI, ADC, and SWI
  Interventions: Device: Cardiac and Brain MRI

INTERVENTIONS:
Device: Cardiac and Brain MRI — A CMR to evaluate for LA and LAA high-risk features on either a 1.5 or 3 Tesla clinical MR scanner will be used. Gadolinium injection will be administered. Gadolinium is a contrast product that helps define areas of fibrosis in the LA.
  High-resolution brain MRI with no contrast will include the following sequences for most accurate assessment of embolic lesions: 3D T1 MPRAGE, 3D FLAIR, DWI, ADC, and SWI

SUMMARY:
Demonstrating the pathophysiological link between Left Atrial (LA) and Left Atrial Appendage (LAA) pathology and embolic strokes in non-Atrial Fibrillation (AF) individuals represents a major advance in stroke prevention strategies. Instead of relying on non-specific criteria for stroke risk assessment, the investigators propose to identify individuals with high-risk of embolic stroke using imaging criteria that reflect the underlying pathophysiology of embolic stroke of cardiac origin. the investigators can therefore lay the groundwork for future anticoagulation strategies for stroke prevention beyond AF.

DETAILED DESCRIPTION:
The investigators propose a cross-sectional cohort study, where individuals with no history of AF and with a Congestive heart failure, Hypertension, Age ≥ 75 years, Diabetes mellitus, Stroke or transient ischemic attack (TIA), Vascular disease, Age 65 to 74 years, Sex category score (CHA2DS2VASC) ≥3, type II diabetes, congestive heart failure or a history of stroke/TIA will be included. Data on demographics, personal health habits, medications, and medical history will be obtained by interviewing participants and reviewing the electronic medical records. All participants will undergo a Cardiac Magnetic Resonance imaging (CMR) to assess for markers of LA and LAA pathology. Markers of LA and LAA pathology that will be studied include: LA fibrosis level, LA functional parameters, LA shape characteristics, and LAA characteristics (including morphology, orifice area and flow velocity). Additionally, all participants will undergo a brain Magnetic Resonance Imaging (MRI) at the same visit to assess for the presence of embolic-appearing brain infarcts, regardless of previous stroke-related symptoms.

The investigators will analyze the association between each cardiac imaging feature and the prevalence of embolic-appearing strokes on brain MRI to determine whether patients with higher LA and LAA remodeled features are more likely to have embolic-appearing brain infarcts on MRI. The LA and LAA pathology imaging features with the strongest statistical association will be used to develop an imaging predictive score capable of identifying patients with the highest risk of embolic stroke.

All brain and cardiac imaging data will be assessed by experienced operators at Tulane Medical Center facilities. Operators analyzing CMR will be blinded to brain MRI results, and operators assessing brain MRI will be blinded to CMR results. The study will include a single center study at Tulane Medical Center and Clinics, with investigators from different medical specialties, and the proper facilities and equipment to conduct the project accurately and safely. The investigators expect a recruitment of 120 subjects over a period of 18 months from both cardiology and neurology clinics to complete the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* 18 Years and older
* No history of atrial fibrillation
* CHA2DS2VASC score ≥3
* History pf type II diabetes
* History of congestive heart failure or a history of transient ischemic attack (TIA)/stroke without an otherwise defined stroke etiology such as large vessel or small vessel disease

Exclusion Criteria:

* History of atrial fibrillation
* Patients who had a clinically symptomatic acute stroke within the last 30-days
* Any health-related gadolinium/MRI contraindication (including previous allergic reaction to Gadolinium, pacemakers, defibrillators, other devices/implants contraindicated for MRI)
* Estimated glomerular filtration rate (eGFR) cutoff in patients with Chronic kidney disease (CKD) where gadolinium cannot be used equals an eGFR <30 ml/min
* Weighing > 300 lbs (as CMR image quality decreases due to increased body mass index)
* Current pregnancy or breastfeeding
* Cognitive impairment preventing the patient from giving an informed consent

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The presence of covert embolic cerebral infarcts | Day1
  The covert embolic cerebral infarcts are defined as the presence of asymptomatic non-lacunar embolic infarct (acute or chronic based on MRI appearance), in the cortex, and juxtacortical regions, and cerebellum. They will be identified using brain MRI.

SECONDARY OUTCOMES:
Number of counts of lacunar covert infracts | Day1
  Covert lacunar infarcts are asymptomatic infarct < 15mm in greatest diameter in subcortical brain regions. They will be identified by size and location using brain MRI images.
Number of counts of lacunar symptomatic infracts | Day1
  Symptomatic lacunar infarcts are symptomatic infarct < 15mm in greatest diameter in subcortical brain regions. They will be identified by size and location using brain MRI images.
Number of counts of embolic symptomatic infracts | Day1
  Symptomatic non-lacunar embolic infarcts are symptomatic infarcts of any size in the cortex or infarcts >15 mm in greatest diameter in subcortical lesions. They will be identified by size and location using brain MRI images.

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Marrouche, MD, Principal Investigator — Tulane School of Medicine
Locations (1):
- Tulane University Medical Center, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Saver JL. CLINICAL PRACTICE. Cryptogenic Stroke. N Engl J Med. 2016 May 26;374(21):2065-74. doi: 10.1056/NEJMcp1503946. No abstract available. PMID 27223148
- [Background] Fanning JP, Wong AA, Fraser JF. The epidemiology of silent brain infarction: a systematic review of population-based cohorts. BMC Med. 2014 Jul 9;12:119. doi: 10.1186/s12916-014-0119-0. PMID 25012298
- [Background] Fanning JP, Wesley AJ, Wong AA, Fraser JF. Emerging spectra of silent brain infarction. Stroke. 2014 Nov;45(11):3461-71. doi: 10.1161/STROKEAHA.114.005919. Epub 2014 Oct 7. No abstract available. PMID 25293663
- [Background] Vermeer SE, Prins ND, den Heijer T, Hofman A, Koudstaal PJ, Breteler MM. Silent brain infarcts and the risk of dementia and cognitive decline. N Engl J Med. 2003 Mar 27;348(13):1215-22. doi: 10.1056/NEJMoa022066. PMID 12660385
- [Background] Gupta A, Giambrone AE, Gialdini G, Finn C, Delgado D, Gutierrez J, Wright C, Beiser AS, Seshadri S, Pandya A, Kamel H. Silent Brain Infarction and Risk of Future Stroke: A Systematic Review and Meta-Analysis. Stroke. 2016 Mar;47(3):719-25. doi: 10.1161/STROKEAHA.115.011889. PMID 26888534
- [Background] Brambatti M, Connolly SJ, Gold MR, Morillo CA, Capucci A, Muto C, Lau CP, Van Gelder IC, Hohnloser SH, Carlson M, Fain E, Nakamya J, Mairesse GH, Halytska M, Deng WQ, Israel CW, Healey JS; ASSERT Investigators. Temporal relationship between subclinical atrial fibrillation and embolic events. Circulation. 2014 May 27;129(21):2094-9. doi: 10.1161/CIRCULATIONAHA.113.007825. Epub 2014 Mar 14. PMID 24633881
- [Background] Daoud EG, Glotzer TV, Wyse DG, Ezekowitz MD, Hilker C, Koehler J, Ziegler PD; TRENDS Investigators. Temporal relationship of atrial tachyarrhythmias, cerebrovascular events, and systemic emboli based on stored device data: a subgroup analysis of TRENDS. Heart Rhythm. 2011 Sep;8(9):1416-23. doi: 10.1016/j.hrthm.2011.04.022. Epub 2011 Apr 23. PMID 21699833
- [Background] Friberg L, Rosenqvist M, Lip GY. Evaluation of risk stratification schemes for ischaemic stroke and bleeding in 182 678 patients with atrial fibrillation: the Swedish Atrial Fibrillation cohort study. Eur Heart J. 2012 Jun;33(12):1500-10. doi: 10.1093/eurheartj/ehr488. Epub 2012 Jan 13. PMID 22246443
- [Background] Fang MC, Go AS, Chang Y, Borowsky L, Pomernacki NK, Singer DE; ATRIA Study Group. Comparison of risk stratification schemes to predict thromboembolism in people with nonvalvular atrial fibrillation. J Am Coll Cardiol. 2008 Feb 26;51(8):810-5. doi: 10.1016/j.jacc.2007.09.065. PMID 18294564
- [Background] Keogh C, Wallace E, Dillon C, Dimitrov BD, Fahey T. Validation of the CHADS2 clinical prediction rule to predict ischaemic stroke. A systematic review and meta-analysis. Thromb Haemost. 2011 Sep;106(3):528-38. doi: 10.1160/TH11-02-0061. Epub 2011 Jul 28. PMID 21800003
- [Background] Marrouche NF, Wilber D, Hindricks G, Jais P, Akoum N, Marchlinski F, Kholmovski E, Burgon N, Hu N, Mont L, Deneke T, Duytschaever M, Neumann T, Mansour M, Mahnkopf C, Herweg B, Daoud E, Wissner E, Bansmann P, Brachmann J. Association of atrial tissue fibrosis identified by delayed enhancement MRI and atrial fibrillation catheter ablation: the DECAAF study. JAMA. 2014 Feb 5;311(5):498-506. doi: 10.1001/jama.2014.3. PMID 24496537
- [Background] Zghaib T, Nazarian S. New Insights Into the Use of Cardiac Magnetic Resonance Imaging to Guide Decision Making in Atrial Fibrillation Management. Can J Cardiol. 2018 Nov;34(11):1461-1470. doi: 10.1016/j.cjca.2018.07.007. Epub 2018 Jul 12. PMID 30297256
- [Background] Bisbal F, Baranchuk A, Braunwald E, Bayes de Luna A, Bayes-Genis A. Atrial Failure as a Clinical Entity: JACC Review Topic of the Week. J Am Coll Cardiol. 2020 Jan 21;75(2):222-232. doi: 10.1016/j.jacc.2019.11.013. PMID 31948652
- [Background] King JB, Azadani PN, Suksaranjit P, Bress AP, Witt DM, Han FT, Chelu MG, Silver MA, Biskupiak J, Wilson BD, Morris AK, Kholmovski EG, Marrouche N. Left Atrial Fibrosis and Risk of Cerebrovascular and Cardiovascular Events in Patients With Atrial Fibrillation. J Am Coll Cardiol. 2017 Sep 12;70(11):1311-1321. doi: 10.1016/j.jacc.2017.07.758. PMID 28882227
- [Background] Daccarett M, Badger TJ, Akoum N, Burgon NS, Mahnkopf C, Vergara G, Kholmovski E, McGann CJ, Parker D, Brachmann J, Macleod RS, Marrouche NF. Association of left atrial fibrosis detected by delayed-enhancement magnetic resonance imaging and the risk of stroke in patients with atrial fibrillation. J Am Coll Cardiol. 2011 Feb 15;57(7):831-8. doi: 10.1016/j.jacc.2010.09.049. PMID 21310320
- [Background] Siebermair J, Suksaranjit P, McGann CJ, Peterson KA, Kheirkhahan M, Baher AA, Damal K, Wakili R, Marrouche NF, Wilson BD. Atrial fibrosis in non-atrial fibrillation individuals and prediction of atrial fibrillation by use of late gadolinium enhancement magnetic resonance imaging. J Cardiovasc Electrophysiol. 2019 Apr;30(4):550-556. doi: 10.1111/jce.13846. Epub 2019 Jan 24. PMID 30661270
- [Background] Habibi M, Zareian M, Ambale Venkatesh B, Samiei S, Imai M, Wu C, Launer LJ, Shea S, Gottesman RF, Heckbert SR, Bluemke DA, Lima JAC. Left Atrial Mechanical Function and Incident Ischemic Cerebrovascular Events Independent of AF: Insights From the MESA Study. JACC Cardiovasc Imaging. 2019 Dec;12(12):2417-2427. doi: 10.1016/j.jcmg.2019.02.021. Epub 2019 Apr 17. PMID 31005519
- [Background] Inoue YY, Alissa A, Khurram IM, Fukumoto K, Habibi M, Venkatesh BA, Zimmerman SL, Nazarian S, Berger RD, Calkins H, Lima JA, Ashikaga H. Quantitative tissue-tracking cardiac magnetic resonance (CMR) of left atrial deformation and the risk of stroke in patients with atrial fibrillation. J Am Heart Assoc. 2015 Apr 27;4(4):e001844. doi: 10.1161/JAHA.115.001844. PMID 25917441
- [Background] Kamel H, Okin PM, Merkler AE, Navi BB, Campion TR, Devereux RB, Diaz I, Weinsaft JW, Kim J. Relationship between left atrial volume and ischemic stroke subtype. Ann Clin Transl Neurol. 2019 Aug;6(8):1480-1486. doi: 10.1002/acn3.50841. Epub 2019 Jul 26. PMID 31402612
- [Background] Al-Saady NM, Obel OA, Camm AJ. Left atrial appendage: structure, function, and role in thromboembolism. Heart. 1999 Nov;82(5):547-54. doi: 10.1136/hrt.82.5.547. PMID 10525506
- [Background] Jeong WK, Choi JH, Son JP, Lee S, Lee MJ, Choe YH, Bang OY. Volume and morphology of left atrial appendage as determinants of stroke subtype in patients with atrial fibrillation. Heart Rhythm. 2016 Apr;13(4):820-7. doi: 10.1016/j.hrthm.2015.12.026. Epub 2015 Dec 18. PMID 26707792
- [Background] Yaghi S, Song C, Gray WA, Furie KL, Elkind MS, Kamel H. Left Atrial Appendage Function and Stroke Risk. Stroke. 2015 Dec;46(12):3554-9. doi: 10.1161/STROKEAHA.115.011273. Epub 2015 Oct 27. No abstract available. PMID 26508750
- [Background] Gaita F, Corsinovi L, Anselmino M, Raimondo C, Pianelli M, Toso E, Bergamasco L, Boffano C, Valentini MC, Cesarani F, Scaglione M. Prevalence of silent cerebral ischemia in paroxysmal and persistent atrial fibrillation and correlation with cognitive function. J Am Coll Cardiol. 2013 Nov 19;62(21):1990-1997. doi: 10.1016/j.jacc.2013.05.074. Epub 2013 Jul 10. PMID 23850917
- [Background] Bokura H, Kobayashi S, Yamaguchi S, Iijima K, Nagai A, Toyoda G, Oguro H, Takahashi K. Silent brain infarction and subcortical white matter lesions increase the risk of stroke and mortality: a prospective cohort study. J Stroke Cerebrovasc Dis. 2006 Mar-Apr;15(2):57-63. doi: 10.1016/j.jstrokecerebrovasdis.2005.11.001. PMID 17904049
- [Background] Debette S, Beiser A, DeCarli C, Au R, Himali JJ, Kelly-Hayes M, Romero JR, Kase CS, Wolf PA, Seshadri S. Association of MRI markers of vascular brain injury with incident stroke, mild cognitive impairment, dementia, and mortality: the Framingham Offspring Study. Stroke. 2010 Apr;41(4):600-6. doi: 10.1161/STROKEAHA.109.570044. Epub 2010 Feb 18. PMID 20167919
- [Background] Gorelick PB, Scuteri A, Black SE, Decarli C, Greenberg SM, Iadecola C, Launer LJ, Laurent S, Lopez OL, Nyenhuis D, Petersen RC, Schneider JA, Tzourio C, Arnett DK, Bennett DA, Chui HC, Higashida RT, Lindquist R, Nilsson PM, Roman GC, Sellke FW, Seshadri S; American Heart Association Stroke Council, Council on Epidemiology and Prevention, Council on Cardiovascular Nursing, Council on Cardiovascular Radiology and Intervention, and Council on Cardiovascular Surgery and Anesthesia. Vascular contributions to cognitive impairment and dementia: a statement for healthcare professionals from the american heart association/american stroke association. Stroke. 2011 Sep;42(9):2672-713. doi: 10.1161/STR.0b013e3182299496. Epub 2011 Jul 21. PMID 21778438
- [Background] Cogswell RJ, Norby FL, Gottesman RF, Chen LY, Solomon S, Shah A, Alonso A. High prevalence of subclinical cerebral infarction in patients with heart failure with preserved ejection fraction. Eur J Heart Fail. 2017 Oct;19(10):1303-1309. doi: 10.1002/ejhf.812. Epub 2017 Jul 24. PMID 28738140
- [Background] Chubb H, Karim R, Roujol S, Nunez-Garcia M, Williams SE, Whitaker J, Harrison J, Butakoff C, Camara O, Chiribiri A, Schaeffter T, Wright M, O'Neill M, Razavi R. The reproducibility of late gadolinium enhancement cardiovascular magnetic resonance imaging of post-ablation atrial scar: a cross-over study. J Cardiovasc Magn Reson. 2018 Mar 19;20(1):21. doi: 10.1186/s12968-018-0438-y. PMID 29554919
- [Background] Margulescu AD, Nunez-Garcia M, Alarcon F, Benito EM, Enomoto N, Cozzari J, Chipa F, Fernandez H, Borras R, Guasch E, Butakoff C, Tolosana JM, Arbelo E, Camara O, Mont L. Reproducibility and accuracy of late gadolinium enhancement cardiac magnetic resonance measurements for the detection of left atrial fibrosis in patients undergoing atrial fibrillation ablation procedures. Europace. 2019 May 1;21(5):724-731. doi: 10.1093/europace/euy314. PMID 30649273
- [Background] Bisbal F, Gomez-Pulido F, Cabanas-Grandio P, Akoum N, Calvo M, Andreu D, Prat-Gonzalez S, Perea RJ, Villuendas R, Berruezo A, Sitges M, Bayes-Genis A, Brugada J, Marrouche NF, Mont L. Left Atrial Geometry Improves Risk Prediction of Thromboembolic Events in Patients With Atrial Fibrillation. J Cardiovasc Electrophysiol. 2016 Jul;27(7):804-10. doi: 10.1111/jce.12978. Epub 2016 May 13. PMID 27027899